CLINICAL TRIAL: NCT03752385
Title: The Effects of Smartphone Use on Physical Activity, Sedentary Behaviour, Sleep, and Well-being
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: University of Prince Edward Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6007767
Record Dates: First submitted 2018-10-12; First posted 2018-11-26 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2018-11

CONDITIONS: Sedentary Lifestyle
Keywords: smartphone; screen time; sedentary behaviour; physical activity; mental health; sleep; adolescents; young adults
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No intervention
- Intervention Group (Experimental): Will cut their smartphone screen time in half, sleep without phone in bedroom, and have a "bedtime" for their phone use.
  Interventions: Behavioral: reducing smartphone screen time

INTERVENTIONS:
Behavioral: reducing smartphone screen time — Cutting average smartphone screen time in half. Sleeping without smartphone in bedroom. Establishing a "bedtime" to stop smartphone screen time.
  Arms: Intervention Group

SUMMARY:
Previous studies suggest that screen use (phones, TV, computers, etc) may negatively impact both sleep and mental health (1-3). The purpose of this study is to determine the impact of reducing smartphone use on sleep, physical activity, sedentary behaviour, and mental health in adolescents and young adults aged 13-25.

DETAILED DESCRIPTION:
Participants will be asked to visit the Active Living Lab on 3 occasions. We expect each visit to take 30-60 minutes.

At baseline, participants will meet with members of the research team to provide informed consent (ages 16+) or parent/guardian consent + participant assent (ages 13-15). Researchers will then record participants' baseline age, gender, height and weight. Participants will then be instructed to download the In The Moment iPhone application which will be used to measure smartphone use. Upon leaving the lab, all participants will be provided with an ActivPAL inclinometer to be worn on the leg, and a Fitbit Flex to be worn on the wrist for 7 days to measure sedentary behaviour, physical activity and sleep.

Following the week of baseline data collection, participants will return to the lab to complete a series of questionnaires focusing on self-reported sedentary behaviour (International Sedentary Assessment Tool, Sedentary Disorder Scale, Social Media Disorder Scale and SHAPES sedentary behaviour questionnaire), physical activity (International Physical Activity Questionnaire), sleep (Pittsburgh Sleep Index), food intake (SHAPES food frequency questionnaire) and mental health (Positive and Negative Affect Schedule and Center for Epidemiologic Studies Depression Scale). At this time participants will also be asked to write down the daily time spent using social media apps (this information can be found under Settings on their iPhone). After completing the questionnaires, participants will be told whether they are in the Intervention or Control groups.

Participants in the intervention group will be asked to restrict their daily smartphone use by 50%, compared to the week of baseline testing. This will be achieved via the OurPact app, which allows the researchers to limit smartphone use to a specific amount of daily use for 7 days (participants will be asked to download and install the app after being told they are in the Intervention group). Once participants have used their allotted daily smartphone time, entertainment apps will not function until the timer is reset the following day (the address book and calling functions are never restricted, so participants will continue to be able to make/receive phone calls, and access their address book at all times). Participants will also be asked to determine a nightly "bedtime", after which their smartphone will be able to make/receive calls, but no other applications will be available. Participants in the intervention group will also be asked to leave their phones outside of their bedroom at night, and will be provided with a digital alarm clock to reduce the use of phones for this purpose.

Participants in the control group will be asked to maintain their typical daily smartphone use for 7 additional days.

After the 7 day intervention/control period, participants will return to the lab to complete the questionnaires for a second time, and to return the Fitbit and inclinometer, and have the apps removed from their phones. Participants in the Intervention group will also be asked to complete a questionnaire on their experience with the intervention, and to provide any additional comments on their experience in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 13 and 25 years of age, own an iPhone, use their phone more than 2 hours/day at baseline and be able to read and write in English.

Exclusion Criteria:

* Outside age limits, does not own an iPhone, cannot read and write in English.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in Positive and Negative Affect | Measured after the first and second week of study.
  Data will be collected using the PANAS scale. Scores for both Positive and Negative Affect range from 10-50, with higher scores representing higher levels of each.
Changes in Depression Symptoms | Measured after the first and second week of study.
  Data will be collected using the CES-D scale. Scores range from 0-60, with higher scores indicating the presence of more symptomatology

SECONDARY OUTCOMES:
Changes in Self-Reported Food Intake | Measured after the first and second week of study.
  Data will be collected using a food frequency questionnaire
Changes in body mass index | Measured after the first and second week of study.
  Calculated using measured height and weight.
Changes in sleep quality and quantity | Measured after the first and second week of study.
  Data will be collected using the Pittsburgh Sleep Quality Index
Changes in Physical Activity | Measured after the first and second week of study.
  Will be assessed via Fitbit
Changes in Sedentary Behaviour | Measured after the first and second week of study.
  Will be measured via ActivPAL inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: Travis Saunders, PHD, Principal Investigator — University of Prince Edward Island
Locations (1):
- University of Prince Edward Island, Charlottetown, Prince Edward Island, Canada